CLINICAL TRIAL: NCT00705666
Title: Real Situation Observational Study of VIRAFERONPEG® in Patients With Chronic Hepatitis C
Brief Title: Treatment of Patients With Chronic Hepatitis C With PegIntron as Monotherapy or in Combination With Ribavirin (Study P04437)(COMPLETED)
Acronym: ADEQUATION
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04437
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepacivirus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PegIntron as monotherapy or in combination with Ribavirin.: Adult participants with chronic hepatitis C treated with PegIntron as monotherapy or in combination with ribavirin.
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b as monotherapy or in combination with ribavirin will be administered according to the products' labeling.
  Other Names: PegIntron
Drug: Ribavirin (SCH 18908) — Peginterferon alfa-2b as monotherapy or in combination with ribavirin will be administered according to the products' labeling.
  Other Names: Rebetol

SUMMARY:
In February 2002, a French Consensus Conference on the management of patients with chronic hepatitis C in France was organized. The jury issued several recommendations on pegylated alpha interferon/ribavirin treatment strategy. Three years after these recommendations, it is of interest to understand the evolution of hepatitis C management in France in real clinical practice. This observational study will permit the identification of patients who are treated and will provide information on the use of PegIntron/ Ribavirin.

DETAILED DESCRIPTION:
To assure a good representation of participants treated for hepatitis C, participants who meet the inclusion criteria will be enrolled on a consecutive basis.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants starting a treatment with PegIntron for the treatment of chronic hepatitis C.

Exclusion Criteria:

* Concomitant participation in a clinical trial for the treatment of hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with chronic hepatitis C treated with PegIntron as monotherapy or in combination with ribavirin at academic centers, clinics, and private practices in France.
Sampling Method: Probability Sample
Enrollment: 789 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PegIntron as Monotherapy or in Combination With Ribavirin
Started | 789
Completed | 450
Not Completed | 339
Not completed — No post-treatment questionnaire | 279
Not completed — Withdrawal by Subject | 21
Not completed — Physician Decision | 7
Not completed — Lost to Follow-up | 5
Not completed — Death | 1
Not completed — Adverse Event | 4
Not completed — Other | 12
Not completed — Other | 2
Not completed — Lack of data | 3
Not completed — Untreated | 5

BASELINE CHARACTERISTICS:
Arm/Group | PegIntron as Monotherapy or in Combination With Ribavirin
Number analyzed (Participants) | 789
Age, Customized [Mean (Standard Deviation); unit: years] | 49 (12.1)
Sex/Gender, Customized [Number; unit: participants] — Gender is provided for the patients that were included in the analysis (781); gender is unknown for the eight (8) participants that were not included in the analysis.
  participants
    Female | 296
    Male | 485
    Unavailable | 8
Region of Enrollment [Number; unit: participants]
  France | 789

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Receiving the Recommended Treatment Duration (24 Weeks for Genotypes 2 and 3 and 48 Weeks for Genotype 1 According to the French 2002 Consensus Meeting).
Time Frame: Physicians will complete a questionnaire at these visits: treatment initiation; 12 and 24 weeks after treatment initiation and 24 weeks after the end of treatment; and 36 and 48 weeks after treatment initiation for participants treated for 48 weeks.
Population: For the 48 week treatment period, the analysis did not separate Genotype 1 (G1) from Genotype 4 (G4) or others. Of the 789 participants, 8 were excluded from analysis (3 for lack of data; 5 because they were untreated).
Measure: Number; unit: Participants
Groups:
- PegIntron as Monotherapy or in Combination With Ribavirin: Adult participants with chronic hepatitis C treated with PegIntron as monotherapy or in combination with ribavirin.
  The recommended treatment duration was 24 weeks for genotypes 2 and 3 and 48 weeks for genotype 1 according to the French 2002 consensus meeting.
  The start and end dates of the treatment were collected in the questionnaire, so the actual treatment duration was calculated for each participant and compared to the theoretical treatment duration reported at Day 0 by the investigators.
Arm/Group | PegIntron as Monotherapy or in Combination With Ribavirin
Number analyzed (Participants) | 781
Participants
  G2, 3 completing 24 weeks of treatment | 160
  G 1, 4, others completing 48 weeks of treatment | 195

ADVERSE EVENTS:
Description: Per protocol, adverse events were not collected; therefore, they were not reported. Serious Adverse Event (SAE) cases were reported by the investigators to the safety department and reported below.
Arm/Group | PegIntron as Monotherapy or in Combination With Ribavirin
Serious Adverse Events (participants affected / at risk) | 66/789
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron as Monotherapy or in Combination With Ribavirin (N=789)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6)
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 1 (1)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 (2)
HYPERSPLENISM (Blood and lymphatic system disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
CARDIAC DISORDER (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
OTOTOXICITY (Ear and labyrinth disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
CONJUNCTIVITIS (Eye disorders) | 1 (1)
IRIDOCYCLITIS (Eye disorders) | 1 (1)
OCULAR HYPERTENSION (Eye disorders) | 1 (1)
RETINAL VEIN OCCLUSION (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4)
ASTHENIA (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1)
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1)
AUTOIMMUNE DISORDER (Immune system disorders) | 1 (1)
INJECTION SITE ABSCESS (Infections and infestations) | 1 (1)
RECTAL ABSCESS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1)
SUPERINFECTION (Infections and infestations) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 (1)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
PATERNAL DRUGS AFFECTING FOETUS (Injury, poisoning and procedural complications) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
BIOPSY LIVER (Investigations) | 1 (1)
ENDOSCOPY GASTROINTESTINAL NORMAL (Investigations) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 (1)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COMA (Nervous system disorders) | 1 (1)
EPILEPSY (Nervous system disorders) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 3 (3)
DELUSION (Psychiatric disorders) | 3 (3)
DEPRESSION (Psychiatric disorders) | 8 (8)
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1)
NERVOUSNESS (Psychiatric disorders) | 1 (1)
PARANOIA (Psychiatric disorders) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 2 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
ALCOHOL DETOXIFICATION (Surgical and medical procedures) | 3 (3)
HOSPITALISATION (Surgical and medical procedures) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any published results concerning the data of the non-interventional study is forbidden. Study data and results are exclusive property of the sponsor.